CLINICAL TRIAL: NCT06627933
Title: Optimization of Management in Patients With Cardiovascular Disease After Lower Limb Joint Replacement
Status: Recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Olga Trushina, Professor, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 11-23
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Thromboembolism; Anticoagulant-induced Bleeding
Keywords: joint replacement; prognosis; anticoagulation regimen; thromboembolism; venous thromboembolism
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low thromboembolic risk
- Moderate thromboembolic risk
- High thromboembolic risk
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: High thromboembolic risk

SUMMARY:
The goal of the study is to evaluate the frequency of cardiovascular and thromboembolic complications in patients with cardiovascular disease after lower limb joint replacement, the influence of known risk factors and strategies for perioperative prevention of thromboembolic complications on the frequency of cardiovascular complications and to develop approaches to optimize antithrombotic prevention tactics.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age older than 18 y.o.
* Cardiovascular disease
* Indications for planned lower limb joint replacement surgery

Exclusion Criteria:

* Pregnancy
* Psychiatric disorders
* Decompensated heart failure or acute heart failure
* Known diagnosis of cancer

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is planned to include 1,000 patients with cardiovascular diseases who undergo routine endoprosthetics of large joints of the lower extremities. During the follow-up, patients will be divided into subgroups depending on the scheme of perioperative prevention of thromboembolic complications and the presence of risk factors. The comparison will be carried out in the appropriate subgroups.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 1 month
  All the cases of major and minor bleeding within 1 month
Bleeding | 3 months
  All the cases of major and minor bleeding within 3 months
Bleeding | 6 months
  All the cases of major and minor bleeding within 6 months
Thromboembolism | 1 month
  All the cases of venous thromboembolism within 1 month
Thromboembolism | 3 months
  All the cases of venous thromboembolism within 3 months
Thromboembolism | 6 months
  All the cases of venous thromboembolism within 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital #1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okisheva EA, Mironova OI, Berdysheva MV, Pyatigorets ES, Krivova NP, Kurnosova AA, Elizarov MP, Smetanin SM, Lychagin AV, Fomin VV. [Relationship between the pain severity, use of non-steroidal anti-inflammatory drugs and blood pressure in elective large joint arthroplasty of the lower extremities]. Ter Arkh. 2023 Nov 3;95(9):751-756. doi: 10.26442/00403660.2023.09.202373. Russian. PMID 38158917
- [Result] Okisheva EA, Trushina OY, Mamaeva MM, Redyanova EA, Zhazhieva AA, Chasova ID, Panferov AS, Bogdanov MM, Lychagin AV, Fomin VV. [Glucose metabolism disorders and hypoglycemic therapy in patients hospitalized for elective lower limb arthroplasty: a prospective, single-center, real-world study]. Ter Arkh. 2024 Jul 30;96(7):659-665. doi: 10.26442/00403660.2024.07.202780. Russian. PMID 39106508